CLINICAL TRIAL: NCT07386626
Title: Study on the Analgesic Effect of Tegileridine Combined With Intercostal Nerve Block After Thoracoscopic Lung Resection
Brief Title: Tegileridine Combined With Intercostal Nerve Block After Thoracoscopic Lung Resection
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, aijun xu, Clinical Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TITL
Record Dates: First submitted 2026-01-22; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Lobectomy
MeSH Terms: interventions — Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sufentanil group (Active Comparator): Administer 0.15 μg/kg (maximum 10 μg) of sufentanil intravenously 40 minutes before the end of surgery, followed by the connection of a sufentanil patient-controlled intravenous analgesia (PCIA)
  Interventions: Procedure: Intercostal Nerve Block; Drug: Sufentanil
- Tegileridine group (Experimental): Administer 0.015 mg/kg (maximum 1mg) of tegileridine intravenously 40 minutes before the end of surgery, followed by the connection of a tegileridine patient-controlled intravenous analgesia (PCIA)
  Interventions: Drug: Tegileridine; Procedure: Intercostal Nerve Block

INTERVENTIONS:
Drug: Tegileridine — Administer 0.015 mg/kg (maximum 1mg) of tegileridine intravenously 40 minutes before the end of surgery, followed by the connection of a tegileridine patient-controlled intravenous analgesia (PCIA)
  Other Names: Tegi
  Arms: Tegileridine group
Procedure: Intercostal Nerve Block — Before closing the chest, the thoracic surgeon injected 3mL of 0.4% ropivacaine into the 4th, 5th, and 6th intercostal spaces through thoracoscopy for intercostal nerve block.
  Other Names: ICNB
Drug: Sufentanil — Administer 0.15 μg/kg (maximum 10 μg) of sufentanil intravenously 40 minutes before the end of surgery, followed by the connection of a sufentanil patient-controlled intravenous analgesia (PCIA)
  Other Names: Sufen
  Arms: sufentanil group

SUMMARY:
Combining tegileridine PCIA with ICNB targeting peripheral nerves, may constitute an ideal analgesic model with complementary advantages. Thus potentially achieving the analgesic goal of "early pain relief, stable throughout the process, and rapid recovery," and may have a positive impact on reducing CPSP.

DETAILED DESCRIPTION:
Combining tegileridine PCIA with ICNB targeting peripheral nerves, may constitute an ideal analgesic model with complementary advantages. ICNB provides rapid and precise incision analgesia in the early postoperative period, effectively blocking the transmission of peripheral nociceptive stimuli to the central nervous system. Tizanidine PCIA, on the other hand, enhances the function of the endogenous descending pain suppression system through its central G protein pathway activation, covering the pain period after the effect of ICNB wears off and components such as visceral referred pain. At the same time, it can effectively reduce side effects such as respiratory depression and nausea/vomiting, thus potentially achieving the analgesic goal of "early pain relief, stable throughout the process, and rapid recovery," and may have a positive impact on reducing CPSP.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 18 to 75 years old;
* Patients undergoing elective thoracoscopic lobectomy or segmentectomy;
* ASA classification levels I-III;
* BMI 18 ~ 30 kg/m2。
* Voluntarily participate and sign an informed consent form.

Exclusion Criteria:

* Patients with preoperative alcohol dependence and long-term use of analgesic drugs are receiving analgesic treatment for other acute and chronic pain;
* Pregnant or lactating women;
* Allergies or other contraindications to the anesthetics, analgesics, and antiemetic drugs used in the study;
* Patients with severe sleep apnea syndrome or acute or severe bronchial asthma;
* Suffering from mental and neurological disorders or cognitive impairment, known or suspected gastrointestinal obstruction, severe liver and kidney dysfunction (Child Pugh score C), chronic obstructive pulmonary disease or severe cardiovascular disease, etc;
* Researchers consider participants who are not suitable to participate in this study and those who refuse to participate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
VAS(Visual Analog Scale） pain score | 48hours
  VAS pain score 0-10, the higher scores mean a worse outcome; Analgesic effect within 48 hours after surgery

SECONDARY OUTCOMES:
Dosage of remedial analgesics | 48hours
  The frequency of remedial analgesia and the total consumption of remedial analgesic drugs
The incidence of ORAEs | 48hours
  The incidence of postoperative opioid related adverse events (ORAEs)

CONTACTS AND LOCATIONS:
Overall Officials: aihua Du, Dr., Study Chair — Tongji Hospital

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) available to other researchers could be requested from the PI Dr. Aijun Xu.